CLINICAL TRIAL: NCT04712188
Title: Shoulder Kinematics and Acute Ultrasonographic Changes in Four Different Stroke Patterns in Manual Wheelchair Users With Spinal Cord Injury
Brief Title: Shoulder Kinematics and Acute Ultrasonographic Changes in Manual Wheelchair Users With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 10
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Traumatic Spinal Cord Injury
Keywords: spinal cord injury; stroke pattern; ultrasonography
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arcing: 10 patients with traumatic spinal cord injury using the "arcing" stroke pattern to propel manual wheelchair
  Interventions: Diagnostic Test: Musculoskeletal ultrasonography; Other: Wheelchair propelling test
- Semicirculer: 10 patients with traumatic spinal cord injury using the "semicirculer" stroke pattern to propel manual wheelchair
  Interventions: Diagnostic Test: Musculoskeletal ultrasonography; Other: Wheelchair propelling test
- Single loop: 10 patients with traumatic spinal cord injury using the "single loop" stroke pattern to propel manual wheelchair
  Interventions: Diagnostic Test: Musculoskeletal ultrasonography; Other: Wheelchair propelling test
- Double loop: 10 patients with traumatic spinal cord injury using the "double loop" stroke pattern to propel manual wheelchair
  Interventions: Diagnostic Test: Musculoskeletal ultrasonography; Other: Wheelchair propelling test

INTERVENTIONS:
Diagnostic Test: Musculoskeletal ultrasonography — The ultrasonographic assesment will be used to examine the supraspinatus tendon thickness, the long head of the biceps brachii tendon thickness and acromio-humeral distance before and after wheelchair propelling test.
Other: Wheelchair propelling test — Participants will use their own wheelchairs with their preferred stroke pattern for 20 minutes at a speed of 1 m / s on a motorized treadmill for a wheelchair propelling test. Wheelchair propelling videos will be recorded during the test. Shoulder kinematics will be analyzed using Kinovea motion analysis software and stoke pattern will be confirmed

SUMMARY:
People who lose function of the lower limb due to spinal cord injury (SCI) need to use their arms for activities of daily life especially during weight-bearing tasks, such as transfers, and manual wheelchair (MWC) propulsion in order to maintain mobility. Persistent use of the upper limbs constitutes biomechanical difficulties, especially in the shoulder joint. The most commonly affected area in the shoulder is supraspinatus and biceps tendon. Four different stoke patterns have been classified in MWC users. Distinct amounts of force may be applied to the shoulder joint during propulsion with different stroke patterns and this can affect the shoulder tendons in different rates. In this study, investigators aimed to evaluate and compare the acute sonographic changes in supraspinatus and biceps tendons after a wheelchair propelling test in MWC users with SCI with different stroke patterns. Also, it is intended to determine the risk factors related to the stroke patterns that may be associated with these sonographic changes.

DETAILED DESCRIPTION:
Fourty male MWC users with SCI were will be divided into 4 groups according to their stroke patterns (arcing, semicirculer, single loop, and double loop). Participants will use their own wheelchairs with their preferred stroke pattern for 20 minutes at a speed of 1 m / s on a motorized treadmill for a wheelchair propelling test. Wheelchair propelling videos will be recorded during the test. Shoulder kinematics will be analyzed using Kinovea motion analysis software and stoke pattern will be confirmed. Ultrasonographic assesment of participants' nondominant shoulder will be performed before and after testing procedure.

ELIGIBILITY:
Inclusion Criteria:

* People with traumatic spinal cord injury
* Age between 18 to 65 years,
* Neurologic injury level at T2 or below, with AIS grade A or B,
* Time since injury at least 6 months,
* Using manual wheelchair as their primary mobility tools

Exclusion Criteria:

* Fractures in nondominant upper limb at any time,
* Shoulder surgery within the past 5 years or corticosteroid injections within the past 3 months to the nondominant shoulder,
* Upper limb pain that restricts propulsion of a manual wheelchair,
* A history of cardiopulmonary problems and degenerative joint diseases

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Fourty male manual wheelchair users with spinal cord injury, will be divided into 4 groups according to their stroke patterns (arcing, semicirculer, single loop, and double loop).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Supraspinatus tendon thickness | Through study completion, an average of 1 month
  Transverse images of the suprasinatus tendon will be performed by using musculoskeletal ultrasonography before and after the wheelchair propelling test
Long head of the biceps tendon thickness | Through study completion, an average of 1 month
  Longitudinal images of the long head of the biceps tendon will be performed by using musculoskeletal ultrasonography before and after the wheelchair propelling test
Acromio-humeral distance | Through study completion, an average of 1 month
  Acromio-humeral distance measurements will be performed by using musculoskeletal ultrasonography before and after the wheelchair propelling test

SECONDARY OUTCOMES:
Shoulder range of motion in the sagittal plane | Through study completion, an average of 1 month
  Shoulder range of motion in the sagittal plane (flexion and extension, degree) will be analyzed using by Kinovea version 0.8.27 motion analysis software.
Contact angle | Through study completion, an average of 1 month
  Contact angle (angle at which the handrim is held, degree) will be analyzed using by Kinovea version 0.8.27 motion analysis software.
Cadence | Through study completion, an average of 1 month
  Cadence (number of strokes per minute, stroke number/minute) will be analyzed using by Kinovea version 0.8.27 motion analysis software.
Push phase | Through study completion, an average of 1 month
  Push phase (time elapsed since the handrim is held until it is released, second) will be analyzed using by Kinovea version 0.8.27 motion analysis software.
Recovery phase | Through study completion, an average of 1 month
  Recovery phase (time elapsed since the handrim is released until it is held again, second) will be analyzed using by Kinovea version 0.8.27 motion analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Korkmaz, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korkmaz N, Yardimci G, Yilmaz B. Temporospatial parameters, shoulder kinematics, and acute tendon changes in four different stroke patterns in male wheelchair users with spinal cord injury. PM R. 2022 Aug;14(8):939-948. doi: 10.1002/pmrj.12733. Epub 2022 Jan 5. PMID 34741794